CLINICAL TRIAL: NCT06969833
Title: Study of Prognostic Factors Associated With Overall Survival in Patients Initially Treated for Advanced Ovarian and/or Peritoneum and/or Fallopian Tubes Carcinoma: Analysis Using a Prospective Clinico-Biological Database
Brief Title: Prospective Clinico-biological Database of Patients With Ovarian and/or Peritoneal and/or Fallopian Tube Carcinoma
Acronym: BCB-OVAIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BCB-OVAIRE-2205
Record Dates: First submitted 2024-09-06; First posted 2025-05-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cancer of the Ovary; Cancer of the Fallopian Tube; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical and Biological Collection (Experimental)
  Interventions: Other: Constitution of a biological collection; Other: Assessment of Quality of Life and level of anxiety/depression

INTERVENTIONS:
Other: Constitution of a biological collection — * Left-over tissue samples (tumor tissue of different nature) frozen and secured in paraffin, and derived from standard care, are collected at study entrance until the end of oncologic treatment.
  * One blood sample of 28mL is collected at time of inclusion
Other: Assessment of Quality of Life and level of anxiety/depression — Questionnaires QLQ-C30, OV-28 and HADS are completed by the patients at inclusion, after 3 and 6 cycles of systemic treatment, and every 3 months up to 2 years after inclusion

SUMMARY:
Cancer of the ovary and/or peritoneum and/or fallopian tube have a very poor prognosis, and require the implementation of collaborative research tools and new innovative therapies. The main objective of this study is to implement prognostic model of overall survival on patients included prospectively as part of the initial treatment of advanced ovarian and/or peritoneum, and/or fallopian tubes carcinoma (this cohort corresponds to the "Turquoise" care pathway of the Oscar Lambret Center) regardless of the treatment carried out,, integrating both patient's and tumor's characteristics. A clinical and biological database is implemented for this purpose.

371 patients will be recruited over a 5-year period at the Oscar Lambret Center.

The active participation of each patient will be 2 years (from the date of inclusion until the end of study participation, defined by the date of the last intervention specific to the research), then the data from standard care and survival data will be collected until the last follow-up of the last patient, 2 years after the last inclusion.

DETAILED DESCRIPTION:
This study is part of the management of patients with advanced ovarian and/or peritoneal carcinoma, and/or fallopian tubes (initial treatment) at the Oscar Lambret Center. Once consent is obtained, registration of patient on the trial is possible during initial care, from diagnosis to the day of surgery.If the diagnosis of advanced invasive ovarian and/or peritoneal and/or fallopian tube carcinoma is finally rejected, patients will be secondarily withdrawn from the study and excluded from analysis.

However, this project differs from standard care with:

* an additional blood sample collected at inclusion (28ml)
* left-over routine samples collected from inclusion until the end of oncologic treatment (tumor samples, ascites, and)
* questionnaires about quality of life (QLQ-C30, QLQ-OV28) and anxiety (HADS) are completed at inclusion, then after 3 and 6 courses of systemic treatment (at the time of laparoscopy or surgery), then every 3 months, up to 2 years after inclusion.
* clinical data are entered into a trial-specific database ; in addition to overall survival, numerous variables will be studied, notably the clinical and socio-economic characteristics of the patients, their planned and effective treatment, the morbidity of treatments, event-free survival, evolution of the quality of life, etc.
* Translational research works will be implemented later on left-over routine samples.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Informed consent warranted
* Patient affiliated to a social security regimen
* Suspected or confirmed diagnosis of advanced and invasive ovarian cancer and/or primary peritoneal cancer and/or fallopian tube cancer (IIB to IV FIGO stages)
* Inclusion during standard care at the Oscar Lambret Centre, from diagnosis to the day of surgery

Exclusion Criteria:

* Patient deprived of liberty or under curatorship or guardianship
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 371 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2032-06-27 (Estimated); Study Completion 2032-06-27 (Estimated)

PRIMARY OUTCOMES:
To identify prognostic factors associated with overall survival on patients included prospectively as part of the initial treatment integrating both patient's and tumor's characteristics, using a multivariate Cox model. | Up to 7 years after the first inclusion
  Overall survival (OS) will defined as the time from the date of histological diagnosis to the date of death whatever the cause.
  Post-relapse OS will be defined as the time from the date of first recurrence to the date of death from any cause.
  The multivariate Cox model will be used to analyze the association of overall survival with prognostic factors:
  * Patient's characteristics: age, weight, body-surface area, Performance status score, ASA score (Physical Status Classification System), antecedents and comorbidities
  * FIGO stage at diagnosis
  * Histological characteristics and histological subtype of tumor: high-grade serous, low-grade serous, endometrioid, clear-cell, mucinous, undifferentiated carcinoma
  * Tumor genetics: HRD or HRP phenotype, methylation, etc.
  * Tumor microenvironment: presence of tumor-infiltrating lymphocytes, presence of tumor-associated Macrophages, and expression of programmed cell death protein-1

SECONDARY OUTCOMES:
To develop a prospective clinico-biological database of patients with advanced ovarian and/or peritoneal and/or fallopian tube carcinoma included during first-line treatment | Up to 7 years after the first inclusion
  * Clinical database created, functional and completed regularly.
  * Biological collection constitued from additional blood samples (1 blood sample of 28ml per patient at the time of inclusion) and from biological extra-samples of standard care (biopsy, ascites)
To develop and validate prognostic models of event-free survival (EFS) on patients included prospectively as part of the initial treatment, integrating both patient's and tumor's characteristics, using a multivariate Cox model | Up to 7 years after the first inclusion
  * Event-free survival will be defined as the time from the date of histological diagnosis to the date of progression, relapse or death from any cause. Patients alive and event-free at the time of the last report will be censored at this date.
  * Post-relapse event-free survival will be defined as the time from the date of the first recurrence to the date of the next event: progression, relapse or death from any cause. Patients who are alive and event-free at the latest will be censored at this date.
  * The multivariate Cox model will be used to analyze the association of EFS with: Patient's characteristics: age, weight, body-surface area, Performance status score, ASA score (Physical Status Classification System), antecedents and comorbidities ; FIGO stage at diagnosis ; Histological characteristics and histological subtype of tumor ; Tumor genetics: HRD or HRP phenotype, methylation, etc. ; Tumor microenvironment: presence of tumor-infiltrating lymphocytes, etc.
To describe both initial characteristics of the patients and their disease characteristics | At baseline
  Clinical data of patients and disease characteristics will be described using traditional methods of descriptive statistics.
  The clinical data include: age, weight, BSA, OMS score, ASA score (Physical Status Classification System), French deprivation index, medical history and comorbidities Disease characteristics include: FIGO stage, ascite, result of biological dosages (CA-125, CA-19.9, inhibine, ACE: carcinoma embryonic antigen), histology, carcinosis index Categorical variables will be presented as frequency and percentage Continuous variables will be presented as median with their extremes or interquartiles, and as mean with standard deviation (the list of data can't be detailed exhaustively in CT.gov).
To describe the therapeutic management of these patients, as planned initially and finally carried out | Up to 7 years after the first inclusion
  The data obtained from standard care will described with usual descriptive statistics:
  * Rate of surgery, complete or not
  * Delay/timing of surgery
  * Rate of systemic treatment: type of chemotherapy and number of courses This multiple measures will be aggregated to mesure the rate of patients receiving the treatment as planned initially, and the rate of patients receiving a treatment different as planned initially.
To describe the morbidity events of first-line treatments | Up to 7 years after the first inclusion
  The number of events will be described by type and by grade (according to NCI-CTCAE V6.0 scale), and for the different phases of treatment (neoadjuvant chemotherapy, surgery, adjuvant chemotherapy).
To describe the distribution of events (recurrence or progression) on patients who have received platinum treatment | Up to 7 years after the first inclusion
  These events will be described according to their time of occurrence in relation to the platinum treatment: during platinum treatment, less than 6 months after the end of platinum treatment, between 6 and 12 months after the end of platinum treatment, after 12 months of platinum treatment
To estimate overall survival (OS) and event-free survival (EFS) of patients | Up to 7 years after the first inclusion
  * Refer to primary outcome for definition and estimation of OS.
  * Refer to secondary outcome linked to prognostic models for definition and estimation of EFS.
To estimate post-relapse overall survival (OS), and post-relapse event-free survival (EFS) of patients | Up to 7 years after the first inclusion
  * Refer to primary outcome for definition and estimation of OS.
  * Refer to secondary outcome linked to prognostic models for definition and estimation of EFS.
To assess the quality of life of patients according to the score calculated with the health-related quality of life questionnaire (QLQ-C30) | At inclusion, after 3 and 6 courses of systemic treatment (up to 3 and 6 months), at the time of surgery, then every 3 months up to 2 years after inclusion
To assess the quality of life of patients according to the score calculated with the ovarian cancer module of the health-related quality of life questionnaire (QLQ-OV28) | At inclusion, after 3 and 6 courses of systemic treatment (up to 3 and 6 months), at the time of surgery, then every 3 months up to 2 years after inclusion
To assess the level of anxiety of patients according to the anxiety score calculated with Hospital Anxiety and Depression scale | At inclusion, after 3 and 6 courses of systemic treatment (up to 3 and 6 months), at the time of surgery, then every 3 months up to 2 years after inclusion
To assess the level of depression of patients according to the depression score calculated with Hospital Anxiety and Depression scale | At inclusion, after 3 and 6 courses of systemic treatment (up to 3 and 6 months), at the time of surgery, then every 3 months up to 2 years after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No